CLINICAL TRIAL: NCT04487236
Title: A Phase 1 Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of ZN-A-1041 Enteric Capsules as a Single Agent or in Combination in Patients With HER2-Positive Advanced Solid Tumors
Brief Title: Trial of ZN-A-1041 Enteric Capsules in Patients With HER2-Positive Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Zanrong Pharma Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ZN-A-1041-101
Record Dates: First submitted 2020-07-10; First posted 2020-07-27 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Advanced Solid Tumors; HER2-positive Breast Cancer
Keywords: Phase 1; Advanced Solid Tumors; HER2-Positive Breast Cancer; Brain metastases
MeSH Terms: conditions — Brain Neoplasms | interventions — BID protein, human; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (11):
- ZN-A-1041 50mg (Experimental): Phase 1a:
  Subjects will be given ZN-A-1041 orally 50mg Bid, for 21days as one cycle
  Interventions: Drug: ZN-A-1041 50mg BID
- ZN-A-1041 100mg (Experimental): Phase 1a:
  Subjects will be given ZN-A-1041 orally 100mg Bid, for 21days as one cycle
  Interventions: Drug: ZN-A-1041 100mg BID
- ZN-A-1041 200mg (Experimental): Phase 1a:
  Subjects will be given ZN-A-1041 orally 200mg Bid, for 21days as one cycle
  Interventions: Drug: ZN-A-1041 200mg BID
- ZN-A-1041 400mg (Experimental): Phase 1a:
  Subjects will be given ZN-A-1041 orally 400mg Bid, for 21days as one cycle
  Interventions: Drug: ZN-A-1041 400mg BID
- ZN-A-1041 600mg (Experimental): Phase 1a:
  Subjects will be given ZN-A-1041 orally 600mg Bid, for 21days as one cycle
  Interventions: Drug: ZN-A-1041 600mg BID
- ZN-A-1041 800mg (Experimental): Phase 1a:
  Subjects will be given ZN-A-1041 orally 800mg Bid, for 21days as one cycle
  Interventions: Drug: ZN-A-1041 800mg BID
- ZN-A-1041 1000mg (Experimental): Phase 1a:
  Subjects will be given ZN-A-1041 orally 1000mg Bid, for 21days as one cycle
  Interventions: Drug: ZN-A-1041 1000mg BID
- ZN-A-1041 level 1+Capecitabine 1000 mg/m2 + Trastuzumab 8 mg/kg iv. First Cycle (Experimental): Phase 1b:
  ZN-A-1041 Level 1 (The previous dose of MTD) to be used in the combination therapy will be determined based on the MTD identified in the Phase 1a study.
  Capecitabine will be given at the dose of 1000 mg/m2, BID (2000 mg/m2/day), during the first 2 weeks of the 21-day treatment cycle.
  Trastuzumab (8 mg/kg in cycle 1 followed by 6 mg/kg beginning in cycle 2, administered as an IV infusion.
  If intolerance, reduce Capecitabine dose to 750 mg/m2 for exploration
  Interventions: Drug: ZN-A-1041 Level 1 +Capecitabine 1000 mg/m2 + Trastuzumab 8 mg/kg iv. First Cycle
- ZN-A-1041 level 2+Capecitabine 1000 mg/m2+ Trastuzumab 8 mg/kg iv. First Cycle (Experimental): Phase 1b:
  ZN-A-1041 Level 2 ( dose of MTD) to be used in the combination therapy will be determined based on the MTD identified in the Phase 1a study.
  Capecitabine will be given at the dose of 1000 mg/m2, BID (2000 mg/m2/day), during the first 2 weeks of the 21-day treatment cycle.
  Trastuzumab (8 mg/kg in cycle 1 followed by 6 mg/kg beginning in cycle 2, administered as an IV infusion.
  If intolerance, reduce Capecitabine dose to 750 mg/m2 for exploration
  Interventions: Drug: ZN-A-1041 Level 2 +Capecitabine 1000 mg/m2 + Trastuzumab 8 mg/kg iv. First Cycle
- ZN-A-1041 MAD+Capecitabine 1000 mg/m2+Trastuzumab 8 mg/kg iv. First Cycle (Experimental): Phase 1b:
  If the MTD is still not reached at the maximum dose level in Phase 1a study, the maximum dose level (MAD) of ZN-A-1041 in Phase 1a will be used in Phase 1b study.
  If intolerance, reduce Capecitabine dose to 750 mg/m2 for exploration
  Interventions: Drug: ZN-A-1041 MAD +Capecitabine 1000 mg/m2 + Trastuzumab 8 mg/kg iv. First Cycle
- ZN-A-1041+Capecitabine+Trastuzumab (Experimental): Phase 1c:
  The combined dose of ZN-A-1041 is based on the recommended combined dose in the Phase 1b and the possible changes in the dosage form and the results of the food effect study, which will be decided by the sponsor and the investigator after discussion
  Interventions: Drug: ZN-A-1041+Capecitabine + Trastuzumab 8 mg/kg iv. First Cycle

INTERVENTIONS:
Drug: ZN-A-1041 50mg BID — Orally 21days for one cycle
  Other Names: ZN-A-1041 Enteric Capsules
  Arms: ZN-A-1041 50mg
Drug: ZN-A-1041 100mg BID — Orally 21days for one cycle
  Other Names: ZN-A-1041 Enteric Capsules
  Arms: ZN-A-1041 100mg
Drug: ZN-A-1041 200mg BID — Orally 21days for one cycle
  Other Names: ZN-A-1041 Enteric Capsules
  Arms: ZN-A-1041 200mg
Drug: ZN-A-1041 400mg BID — Orally 21days for one cycle
  Other Names: ZN-A-1041 Enteric Capsules
  Arms: ZN-A-1041 400mg
Drug: ZN-A-1041 600mg BID — Orally 21days for one cycle
  Other Names: ZN-A-1041 Enteric Capsules
  Arms: ZN-A-1041 600mg
Drug: ZN-A-1041 800mg BID — Orally 21days for one cycle
  Other Names: ZN-A-1041 Enteric Capsules
  Arms: ZN-A-1041 800mg
Drug: ZN-A-1041 1000mg BID — Orally 21days for one cycle
  Other Names: ZN-A-1041 Enteric Capsules
  Arms: ZN-A-1041 1000mg
Drug: ZN-A-1041 Level 1 +Capecitabine 1000 mg/m2 + Trastuzumab 8 mg/kg iv. First Cycle — ZN-A-1041 level 1 BID; Capecitabine 1000 mg/m2 BID Trastuzumab 8 mg/kg iv. First Cycle
  Other Names: ZN-A-1041 Enteric Capsules
  Arms: ZN-A-1041 level 1+Capecitabine 1000 mg/m2 + Trastuzumab 8 mg/kg iv. First Cycle
Drug: ZN-A-1041 Level 2 +Capecitabine 1000 mg/m2 + Trastuzumab 8 mg/kg iv. First Cycle — ZN-A-1041 level 2 BID; Capecitabine 1000 mg/m2 BID Trastuzumab 8 mg/kg iv. First Cycle
  Other Names: ZN-A-1041 Enteric Capsules
  Arms: ZN-A-1041 level 2+Capecitabine 1000 mg/m2+ Trastuzumab 8 mg/kg iv. First Cycle
Drug: ZN-A-1041 MAD +Capecitabine 1000 mg/m2 + Trastuzumab 8 mg/kg iv. First Cycle — ZN-A-1041 MAD BID; Capecitabine 1000 mg/m2 BID Trastuzumab 8 mg/kg iv. First Cycle
  Other Names: ZN-A-1041 Enteric Capsules
  Arms: ZN-A-1041 MAD+Capecitabine 1000 mg/m2+Trastuzumab 8 mg/kg iv. First Cycle
Drug: ZN-A-1041+Capecitabine + Trastuzumab 8 mg/kg iv. First Cycle — Base on 1b ZN-A-1041 dose Base on 1b Capecitabine dose Base on 1b Trastuzumab dose
  Other Names: ZN-A-1041 Enteric Capsules
  Arms: ZN-A-1041+Capecitabine+Trastuzumab

SUMMARY:
This will be a phase 1, multicenter, open-label trial to evaluate the safety, tolerability, PK and efficacy of ZN-A-1041 as a monotherapy or in combination in patients with HER2-positive advanced solid tumors.

The study will consist of three phases: phase 1a (dose escalation with ZN-A-1041 monotherapy), phase 1b (dose escalation with ZN-A-1041 in combination with Capecitabine and Trastuzumab) and phase 1c (dose expansion with ZN-A-1041 in combination with Capecitabine and Trastuzumab).

DETAILED DESCRIPTION:
Phase 1a of the study will adopt the "modified 3+3" dose escalation design with a total of 7 planned dose levels. Patients with HER2-positive advanced solid tumor (including those with brain metastases) will be enrolled to receive a single-dose administration of ZN-A-1041 followed by multiple-dose administration of ZN-A-1041.

Phase 1b of the study will adopt the "traditional 3+3" dose escalation design. In phase 1b, patients with HER2-positive advanced breast cancer (including those with brain metastases) will be enrolled to receive multiple doses of ZN-A-1041 in combination with Capecitabine and Trastuzumab.

In phase 1c patients with HER2-positive breast cancer with brain metastases were planned to be enrolled to receive ZN-A-1041 in combination with Capecitabine and Trastuzumab The dose levels will be determined based on the recommended doses obtained from the Phase 1b study, and the possible changes in the dosage form and the food effect study, which will be decided by the sponsor and the investigator after discussion.

Each phase of the study includes a screening period, a treatment period and a follow-up period. During the trial, the safety, tolerability, PK and efficacy data of ZN-A-1041 as monotherapy and in combination with Capecitabine and Trastuzumab in the subjects will be collected and analyzed, thereby providing RP2D for the subsequent clinical trials.

ELIGIBILITY:
Key inclusion criteria:

11. ECOG performance status of 0 to 1 2. HER2-positive is defined as Immunohistochemistry (IHC) (++) and Fluorescence In Situ Hybridization (FISH) positive, or IHC (+++).

3. Phase 1a study will enroll patients with unresectable or metastatic HER2-positive advanced solid tumor; Phase 1b study will enroll patients with unresectable locally-advanced or metastatic HER2+ breast cancer.

i. For patients who have no brain metastases, the following criteria should be met:

1. Patients should be relapsed or refractory to existing therapy(ies) or have been intolerant of such therapies
2. Have at least one extracranial measurable lesion by RECIST v1. 1 ii. For patients with brain metastasis, the following criteria should be met:

1) Have received prior treatment or patient declined the above treatment; 2) Patients with HER2-positive gastric cancer must have previously received Trastuzumab 3) Do not require immediate local treatment during the trial period, and meet either of the following two criteria:

1. For patients who have received previous local treatment (surgery, whole brain radiotherapy (WBRT) and stereotactic radiosurgery (SRS)) for brain metastases, stable or progression of intracranial lesions is required. Interval from prior local therapy could be 3 weeks from WBRT and 2 weeks from SRS.
2. Symptomatic or not, patient has not received previous local treatment (surgery or radiotherapy) for brain metastases as long as no local therapy is needed during the trial period.

iii. In Phase 1a, for patients who have received previous tyrosine kinase inhibitor (TKI) treatment, chemotherapy, antibody, or antibody-drug conjugate (ADC), the interval between the last treatment and the first administration of the study drug in this trial should be at least 2 weeks. In Phase 1b, for patients who have received previous trastuzumab or other antibodies, the interval between the last treatment and the first administration of the study drug in this trial should be at least 3 weeks.

4. Phase 1c study will enroll patients with unresectable locally-advanced or metastatic HER2+ breast cancer with brain metastases.

i. For patients with brain metastasis, patients do not require immediate local treatment during the trial period, and meet either of the following two criteria:

1. For patients who have received previous local treatment (surgery, whole brain radiotherapy (WBRT) and stereotactic radiosurgery (SRS)) for brain metastases, stable or progression of intracranial lesions is required. Interval from prior local therapy could be 3 weeks from WBRT, 2 weeks from SRS and 4 weeks from surgery
2. Symptomatic or not, patient has not received previous local treatment (surgery or radiotherapy) for brain metastases as long as no local therapy is needed during the trial period
3. Have at least one measurable lesion and is suitable for accurate repeated assessable by RECIST 1.1, and the patient has an imaging-diagnosable intracranial lesion;
4. Patients should not include suspected or confirmed meningeal metastases;
5. The patient had no disease progression with previous 12 weeks' capecitabine therapy;
6. No capecitabine therapy within 6 months;
7. Patient should not previously treat with a tyrosine kinase inhibitor (TKI). Previous treatment with trastuzumab or other antibodies should be at least 3 weeks apart from the first treatment

Key exclusion criteria:

1. Subjects who have participated in any clinical study or received any clinical study drug within 4 weeks prior to the first administration
2. There is evidence that other primary tumors are present at the same time;
3. Previous cumulative dose of doxorubicin exceeds 360mg/m2 or its equivalent dose of similar drugs;
4. CNS Exclusion - Based on screening brain MRI and clinical assessment

   1. Progressive neurologic impairment or increased intracranial pressure (including nausea, vomiting, blurred vision, headache, epilepsy, etc.)
   2. Any intracranial lesion thought to require immediate local therapy
   3. Require antiepileptic treatment (except for these patients with stable seizures require continuous Levetiracetam therapy).
   4. Ongoing use of systemic corticosteroids for control of symptoms of brain metastases at a total daily dose of > 2 mg of dexamethasone (or equivalent)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2024-04-16 (Actual); Study Completion 2025-04-16 (Actual)

PRIMARY OUTCOMES:
The safety/tolerability of ZN-A-1041 as a monotherapy on Phase 1a | 23days
  Dose at which no more than one out of six patient at the same dose level experiences a probable drug-related dose limiting toxicity.
The safety/tolerability of ZN-A-1041 in combination with Capecitabine and Trastuzumab in Phase 1b | 21days
  Dose at which no more than one out of six patient at the same dose level experiences a probable drug-related dose limiting toxicity.
The safety of ZN-A-1041 in combination with Capecitabine and Trastuzumab in Phase 1c | through study completion, an average of 3 year
  To evaluate the safety of ZN-A-1041 in combination with Capecitabine in patients on the RP2D Dose

SECONDARY OUTCOMES:
Plasma Level of ZN-A-1041 and its major metabolites on phase 1a,phase 1b and 1c | From baseline to Day 8
  To assess the AUC of ZN-A-1041 and its major metabolites;
Plasma Level of ZN-A-1041 and its major metabolites on Phase 1a,phase 1 b and 1c | From baseline to Day 8
  To assess the Cmax of ZN-A-1041 and its major metabolites;
Plasma level of ZN-A-1041 and its main metabolites Phase 1a,phase 1b and 1c | From baseline to Day 8
  To assess the Tmax of ZN-A-1041 and its major metabolites;
The preliminary efficacy of ZN-A-1041 as a monotherapy or combination in Phase 1a,phase 1b and 1c | through study completion, an average of 3 year
  overall Response Rate (ORR);Progression free survival(PFS)

CONTACTS AND LOCATIONS:
Overall Officials: Fei Ma, MD, Principal Investigator — Cancer Hospital, Chinese Academy of Medical Sciences, Peking Union Medical College
Locations (1):
- Cancer hospital Chinese academy of medical sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No